CLINICAL TRIAL: NCT04740437
Title: Interest of Systematic PPI Therapy After POEM vs Symptomatic Use of PPI Therapy in Prevention of Gastroesophageal Reflux Disease After POEM for Esophageal Achalasia. A Comparative Retrospective Analysis.
Brief Title: Systematic IPP VS Symptomatic IPP in GERD Prevention After POEM for Achalasia. . A Comparative Retrospective Analysis
Acronym: IPPOEM-Retro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0064
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Achalasia; Gastroesophageal Reflux
Keywords: GERD; POEM; Achalasia; PPI; Esophagitis
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux; Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
POEM is a minimally invasive endoscopic therapy that is highly efficacy in the treatment of achalasia of any type. POEM has an increased risk of GERD. Systematic PPI therapy has never been studied for the prevention of post-POEM GERD.

The investigators wish to retrospectively compare patients who have received routine PPI therapy vs. patients who don't.

ELIGIBILITY:
Inclusion criteria:

* > 18 years old
* Consent given
* Achalasia all types with eckhardt score > 3

Exclusion criteria:

* Patient who is a minor or under judicial protection
* Pregnant or breastfeeding woman
* Contraindication to PPIs
* Carrier of mediastinal and exogastric neoplasia
* Patient on PPIs prior to the procedure for indication that does not allow for their discontinuation
* Peptic esophagitis (Grade B, C or D) before or at the time of the procedure
* Previous treatment with Heller myotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included from several French university hospitals that have POEM as a treatment for esophageal achalasia and which routinely perform an endoscopic evaluation of esophagitis between 6 to 9 months after the POEM.
  Data collection will be retrospective from patient records at each center.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Esophagitis | 1 day
  Number of Esophagitis

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Debourdeau, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
nc